CLINICAL TRIAL: NCT01879670
Title: Partial Left Ventricular Support in Advanced Heart Failure
Status: Terminated | Type: Observational
Why Stopped: Withdrawal of CircuLite Synergy from clinical use
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: 2012HSB002B; FS/13/34/30173 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2013-06-11; First posted 2013-06-18 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure; Heart-Assist Devices
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Synergy: Patients in the Synergy group will have severe advanced heart failure (see inclusion criteria) and will have been selected by their clinical team for implantation of a CircuLite Synergy left ventricular assist device.
  Interventions: Device: CircuLite Synergy left ventricular assist device
- Control: Patients in the Synergy group will have severe advanced heart failure (see inclusion criteria) and will have been selected by their clinical team to continue current optimal medical and device therapy.

INTERVENTIONS:
Device: CircuLite Synergy left ventricular assist device
  Other Names: CircuLite Synergy circulatory assist device; SIK 100
  Groups: Synergy

SUMMARY:
Heart failure is a common condition, and the number of people with advanced disease continues to increase. We need new treatments that improve patients' symptoms and extend life. Recently the new CircuLite Synergy pump has come into use. It is the smallest pump manufactured to date and does not cover the full work of the heart, instead providing "partial" support. One interesting thing about this is that taking some strain off the heart might allow the muscle to repair and rebuild its own strength. This process is called reverse remodelling, and is the topic of this research. Our hypothesis is that "partial" support improves patients' symptoms and causes improvement in heart muscle function. We also want to examine the best techniques for assessing this, including new scanning and molecular tests, and study some practical aspects of the pump to do with blood clotting.

DETAILED DESCRIPTION:
The CircuLite Synergy pump is a new minimally-invasive partial support left ventricular assist device (LVAD) that pumps blood from the left atrium to the right subclavian artery. Ex vivo pilot data suggests that the Synergy pump induces structural reverse remodelling, which proposes the Synergy device as a new disease-modifying therapy. We will assess whether the Synergy pump facilitates functional, structural and molecular LV reverse remodelling in vivo; assess how this can be determined and predicted by analysis of circulating micro RNA profiles and specific echocardiographic parameters; and evaluate the haematological abnormalities associated with this new LVAD.

We will address these questions with a prospective, observational study comparing patients implanted with the Synergy device with matched heart failure controls. The two study centres will be Royal Brompton & Harefield NHS Foundation Trust (Harefield Hospital) and University Hospitals Leuven, Belgium. We will recruit a total of 64 patients. The primary outcome will be change in peak VO2 at 6 months. Secondary outcomes will include functional parameters, profiling of circulating microRNA, multimodal echocardiographic assessment and comprehensive assessment of platelet activation and coagulopathy.

We will quantify the LV reverse remodelling associated with partial support; define new echo and microRNA markers of reverse remodelling for clinical use, with insights into underlying pathophysiology; and describe the haematological profile of these patients to guide future antiplatelet and anticoagulant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischaemic or dilated cardiomyopathy aged 18 to 80 years.
* Symptoms categorised by INTERMACS (Interagency Registry for Mechanically Assisted Circulatory Support) at level 3-6 despite optimal tolerated medical therapy. Practically this includes patients who are in hospital or managing at home with substantial dependence on hospital care.
* Peak VO2 <15ml/kg/min with respiratory exchange ratio>1 on cardiopulmonary exercise testing OR a 6-minute walking distance <300m OR inability to perform an exercise test due to the severity of heart failure.
* Informed consent obtained prior to entering the study.

Exclusion Criteria:

* Cause of heart failure due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis, or active myocarditis
* Body surface area <1.2M2 or >2.3M2, or body mass index >32 kg/M2.
* Severe chronic obstructive pulmonary disease as evidenced by forced expiratory volume in 1 second <50% of predicted.
* History of pulmonary hypertension with maintained pulmonary vascular resistance measured > 4 Wood units or transpulmonary gradient >14mmHg.
* Pregnancy.
* Evidence of intrinsic hepatic disease defined as liver enzyme levels > 5 times the upper limit of normal within 4 days before enrolment, severe liver dysfunction, cirrhosis or portal hypertension.
* Occurrence of stroke within 90 days before enrolment.
* Impairment of cognitive function or presence of any form of irreversible dementia.
* Recent history of psychiatric disease (including severe drug or alcohol abuse) that is likely to impair compliance with the study protocol.
* Platelet count <50 x103mm3 within 24 hours before enrolment.
* Creatinine clearance < 30ml/min.
* High probability of non-compliance.
* The patient is deemed unsuitable by the clinical team for other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from advanced heart failure clinics at two tertiary heart hospitals with large cardiac transplantation and mechanical circulatory support programmes.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in maximal aerobic exercise capacity (peak VO2) | 6 months

SECONDARY OUTCOMES:
Change in 6-minute walk distance | 6 months
Change in New York Heart Association (NYHA) functional class | 6 months
Change in B-type natriuretic peptide | 6 months
Change in ventricular dimensions as measured by echocardiography | 6 months
Change in ventricular strain as measured by echocardiography | 6 months
Change in circulating microRNA expression profile | 6 months
Change in ventilatory equivalent for carbon dioxide (VE/VCO2) slope | 6 months
Change in haemodynamic parameters at right heart catheterisation | 6 months
Change in quality of life score | 6 months
Accumulated days of hospital inpatient stay due to cardiovascular reasons | 6 months
Incidence of significant haematological derangements | 6 months
Number of participants suffering adverse events | 6 months
  'Adverse events' are defined as major bleeding, thromboembolism, stroke, infection, perioperative complications, right ventricular failure, device-related morbidity and device failure.

CONTACTS AND LOCATIONS:
Overall Officials: John R Pepper, FRCS, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust and Imperial College London
Locations (2):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Royal Brompton & Harefield NHS Foundation Trust, London, United Kingdom

REFERENCES:
- See also: Royal Brompton & Harefield NHS Foundation Trust — http://www.rbht.nhs.uk/
- See also: Universitaire Ziekenhuizen Leuven — http://www.uzleuven.be/en